CLINICAL TRIAL: NCT03641170
Title: The Acute Effect of Physical Activity on Postprandial Blood Glucose in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Diet study
Record Dates: First submitted 2018-04-09; First posted 2018-08-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-01

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention (Experimental): Fixed diet and physical activity.
  Interventions: Behavioral: Physical activity; Other: Fixed diet.
- Control intervention (Other): Fixed diet and inactivity.
  Interventions: Behavioral: Inactivity; Other: Fixed diet.

INTERVENTIONS:
Behavioral: Physical activity — Interval walking performed after each main meal.
  Arms: Experimental intervention
Behavioral: Inactivity — Inactivity after each main meal.
  Arms: Control intervention
Other: Fixed diet. — Participants will receive a fixed diet through out the intervention period and control period.

SUMMARY:
The aim of the project is to investigate the acute effect of exercise on blood glucose after food consumption. Thereby the investigators wish to achieve knowledge that can improve prevention and treatment of gestational overweight and gestational diabetes mellitus (GDM). This will prevent serious complications during pregnancy and birth, but also long term complications like type 2 diabetes mellitus (T2DM) for both the mother and the offspring.

Inclusion will be 60 pregnant women divided into three groups - normal weight, overweight and obese and women with gestational diabetes. Participants will receive a fixed diet and go through an intervention period with physical activity immediately after each main meal and a control period with inactivity after the meals. Blood glucose will be the main outcome.

DETAILED DESCRIPTION:
Design: Crossover controlled study. Cases: 60 pregnant women recruited at the Department of Obstetrics and Gynecology, Aarhus University Hospital (AUH). Subjects will receive both written and oral information before entering the trial. According to their prepregnancy BMI, subjects will be recruited for three different groups: i) normal weight (BMI 18,5-24,9), ii) overweight and obese (BMI ≥ 25) and iii) GDM. 20 women in each group. Group i and ii will be recruited at the routine ultrasound scan at gestational week 19. Group iii will be recruited after the Oral Glucose Tolerance Test (OGTT) that diagnoses gestational diabetes mellitus. The routine OGTT is done at gestational week 28. When diagnosed with GDM the women are referred to Department of Obstetrics and Gynecology, AUH, and the investigators will recruit participants from here. Participants will be examined during gestational week 30-34 where insulin resistance peaks during pregnancy.

Intervention: Participants will receive a fixed diet for a total of 8 days. The 8 days of fixed diet are split into a 4 days intervention period and a 4 days control period separated by two days of regular food intake. The two days of regular food intake will function as a "wash out period" to avoid carry over effect. During the 4 days intervention period the participants will perform 30 minutes of interval walking immediately after each main meal. The interval walking consists of alternating fast and slow intervals (3 minutes each) aiming at > 70% and < 40% of peak energy expenditure measured by the Sensewear Armband. During the 4 days control period the participants will be normally active, not performing any set physical activity. Participants will be randomized to the order of the two periods.

Study variables: Fasting blood samples will be taken on the first day of both the intervention and control period and on the morning after the last day of each period. Blood samples will be analyzed for blood glucose, HbA1c, C-peptide and lipid profile (triglycerides, HDL and LDL).

During the entire experimental period, movement data will be collected using the Sensewear Armband. Blood glucose will be monitored continuously using the IPro2 Continuous Glucose Monitor (CGM) from Medtronic.

The diet will consist of three main meals and three snacks and will be calculated to match their metabolic need. The calculations will be done by a nutrition specialist and will include weight, height, BMI and energy need during 3rd trimester pregnancy.

Data on demography, family history of diabetes, prepregnancy BMI, gestational weight gain and complications during pregnancy are collected from medical records of the patients and their offspring.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over age of 18
* according to each group: BMI: 18,5-24,9; BMI: >25; women with GDM.

Exclusion Criteria:

* women with a physical disability that affects their movement will be excluded from the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Through intervention periods of 4 days.
  Differences in blood glucose between experimental intervention (physical activity) and control intervention (inactivity).

CONTACTS AND LOCATIONS:
Overall Officials: Per Ovesen, MD, Prof., Study Director — Aarhus University Hospital / University of Aarhus
Locations (1):
- Department of Obstetrics and Gynecology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen MB, Fuglsang J, Ostenfeld EB, Poulsen CW, Daugaard M, Ovesen PG. Postprandial interval walking-effect on blood glucose in pregnant women with gestational diabetes. Am J Obstet Gynecol MFM. 2021 Nov;3(6):100440. doi: 10.1016/j.ajogmf.2021.100440. Epub 2021 Jun 30. PMID 34216833